CLINICAL TRIAL: NCT01873794
Title: Treating Cancer-Related Fatigue Through Systematic Light Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of California, San Diego (Other); Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GCO 10-0864; 5R21CA158954 (NIH); HSM#11-01032
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Hematopoietic Stem Cell Transplantation; Breast Cancer; Fatigue; Mild Cognitive Impairment; Light; Quality of Life; Sleep
Keywords: Fatigue; Sleep; Quality of life; Cancer; Light
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Cognitive Dysfunction; Neoplasms | interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright white light (Active Comparator): using systematic light exposure (SLE), consisting of a daily 30-minute exposure to as much as 10,000 lux of light from a commercially available light box
  Interventions: Device: Bright white light
- Dim red light (Active Comparator): using systematic light exposure (SLE), consisting of a daily 30-minute exposure to as much as 10,000 lux of light from a commercially available light box
  Interventions: Device: Dim red light

INTERVENTIONS:
Device: Bright white light
  Other Names: Light Box; Litebook
  Arms: Bright white light
Device: Dim red light
  Other Names: Light Box; Litebook
  Arms: Dim red light

SUMMARY:
Cancer related fatigue (CRF) - a persistent sense of exhaustion related to cancer or cancer treatment - can severely interfere with activities of daily living, and has even been reported to be a factor in patient requests for hastened death. CRF can represent a serious clinical problem years after all treatment has ended. There is currently no effective treatment for CRF. The purpose of this study is to investigate whether systematic exposure to light (from a commercially available Litebook) reduces CRF or other symptoms.

DETAILED DESCRIPTION:
Cancer related fatigue (CRF) - a persistent sense of exhaustion related to cancer or cancer treatment - can severely interfere with activities of daily living, and has even been reported to be a factor in patient requests for hastened death. CRF can represent a serious clinical problem years after all treatment has ended. In our research with cancer survivors 1 to 3 years after completion of hematopoietic stem cell transplant (HSCT), 40% of those we interviewed reported that CRF was a major obstacle to the resumption of usual activities. Despite its impact on quality of life, CRF is under-reported, under-diagnosed, and under-treated.

A variety of pharmacologic agents have been studied to treat CRF, but there is insufficient evidence to recommend their use. The most promising non-pharmacologic interventions -- exercise and cognitive-behavior therapy (CBT) -- have shown equally modest effects. The proposed study focuses on a promising new intervention for CRF, using systematic light exposure (SLE), consisting of a daily 30-minute exposure to as much as 10,000 lux of light from a commercially available light box. Study collaborator, Ancoli-Israel and her colleagues have successfully piloted this line of research with breast cancer patients undergoing chemotherapy.

The goal of this study will be to assess the effect of SLE on long-term HSCT and breast cancer survivors, and to determine the feasibility and acceptability of SLE as an intervention for CRF. The approach will be informed by the procedures that Ancoli-Israel and her colleagues developed for their research on SLE treatment for breast cancer chemotherapy, as well as by Redd's studies of CBT to treat adjustment disorders in survivors of HSCT. The study arms will test the efficacy of two different types of light treatment, bright white light and dim red light. Outcomes will be assessed through standardized measures of CRF, sleep quality, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* With a history of HSCT as treatment for hematological malignancies and related diseases and who are up to 3.5 years post-transplant; OR
* Who are up to three and a half years post completion of chemotherapy OR chemotherapy and radiation for breast cancer with a curative intent;

AND:

* With a score equal to or less than 33 on the FACIT-Fatigue scale (see below) and no pre-existing anemia (Hb<10gm/dl); or a score equal to or greater than 43 on the Cognitive Failures Questionnaire
* Who are currently over age 18 and at least age 16 at the time of HSCT or time of breast cancer treatment

Exclusion Criteria:

* Under age 18;
* Pregnancy;
* Confounding underlying medical illnesses;
* History of mania (which is a contra-indication for light treatment) or current clinical depression;
* And any other physical or psychological impairments including a sleep disorder diagnosis which would limit participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
FACIT-Fatigue Scale | Baseline
  A list of statements that patients with cancer have said about their fatigue will be read. Subjects will mark on a 5-point scale how often they have felt each statement over the last 7 days. Measured at baseline, second week of light box use, fourth (last) week of light box use, three weeks post completion of light box use
FACIT-Fatigue Scale | at 4 weeks
  A list of statements that patients with cancer have said about their fatigue will be read. Subjects will mark on a 5-point scale how often they have felt each statement over the last 7 days.
FACIT-Fatigue Scale | at 3 months follow up
  A list of statements that patients with cancer have said about their fatigue will be read. Subjects will mark on a 5-point scale how often they have felt each statement over the last 7 days.

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index | Baseline
  The validity of the instrument is based on its ability to discriminate patients (those having either sleep problems and/or depressive symptoms) from controls (healthy participants without sleep complaints). Baseline, second week of light box use, fourth (last) week of light box use, three weeks post completion of light box use
The Pittsburgh Sleep Quality Index | at 4 weeks
  The validity of the instrument is based on its ability to discriminate patients (those having either sleep problems and/or depressive symptoms) from controls (healthy participants without sleep complaints).
The Pittsburgh Sleep Quality Index | at 3 months follow up
  The validity of the instrument is based on its ability to discriminate patients (those having either sleep problems and/or depressive symptoms) from controls (healthy participants without sleep complaints.
SF-36 Scale | Baseline
  Quality of life will be assessed using the SF-36 scale. The SF-36 is a multi-purpose, short form health survey consisting of 36 questions.
SF-36 Scale | at 4 weeks
  Quality of life will be assessed using the SF-36 scale. The SF-36 is a multi-purpose, short form health survey consisting of 36 questions.
SF-36 Scale | at 3 months follow up
  Quality of life will be assessed using the SF-36 scale. The SF-36 is a multi-purpose, short form health survey consisting of 36 questions.
CNS-Vital Signs | Baseline
  Objective cognitive function will be assessed using CNS-Vital Signs, a reliable and valid computer-administered cognitive assessment battery that consists of 7 cognitive tests.
CNS-Vital Signs | at 4 weeks
  Objective cognitive function will be assessed using CNS-Vital Signs, a reliable and valid computer-administered cognitive assessment battery that consists of 7 cognitive tests.
CNS-Vital Signs | at 3 months follow up
  Objective cognitive function will be assessed using CNS-Vital Signs, a reliable and valid computer-administered cognitive assessment battery that consists of 7 cognitive tests.
The Cognitive Failures Questionnaire | Baseline
  A 25-item self-report measure of cognitive difficulties in everyday life using a 5-point Likert scale.
The Cognitive Failures Questionnaire | at 4 weeks
  A 25-item self-report measure of cognitive difficulties in everyday life using a 5-point Likert scale.
The Cognitive Failures Questionnaire | at 3 months follow up
  A 25-item self-report measure of cognitive difficulties in everyday life using a 5-point Likert scale.
Brief Symptom Inventory-18 | Baseline
  Used to assess psychological distress. A list of health problems and complaints that people sometimes experience are listed.
Brief Symptom Inventory-18 | at 4 weeks
  Used to assess psychological distress. A list of health problems and complaints that people sometimes experience are listed.
Brief Symptom Inventory-18 | at 3 months follow up
  Used to assess psychological distress. A list of health problems and complaints that people sometimes experience are listed.
Actiwatch Spectrum | Baseline
  Sleep/wake activity is measured using an actigraph which records physical movement and detects light. The Actiwatch is worn for 72 consecutive hours.
Actiwatch Spectrum | at 4 weeks
  Sleep/wake activity is measured using an actigraph which records physical movement and detects light. The Actiwatch is worn for 72 consecutive hours.
Actiwatch Spectrum | at 3 months follow up
  Sleep/wake activity is measured using an actigraph which records physical movement and detects light. The Actiwatch is worn for 72 consecutive hours.

CONTACTS AND LOCATIONS:
Overall Officials: William H Redd, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Derived] Wu LM, Amidi A, Valdimarsdottir H, Ancoli-Israel S, Liu L, Winkel G, Byrne EE, Sefair AV, Vega A, Bovbjerg K, Redd WH. The Effect of Systematic Light Exposure on Sleep in a Mixed Group of Fatigued Cancer Survivors. J Clin Sleep Med. 2018 Jan 15;14(1):31-39. doi: 10.5664/jcsm.6874. PMID 29198295